CLINICAL TRIAL: NCT06530342
Title: Determination of the Effect of Hamstring Muscle Length on Lunge Distance in Fencing Athletes
Brief Title: Effect of Hamstring Muscle Length on Lunge Distance in Fencing Athletes
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Other Study IDs: 28.07.2024-EÜ
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fencing Sword Branch Athletes: 20 volunteer sword fencing athletes who are licensed by the Anatolian Archery and Fencing Club and meet our inclusion criteria.
  Interventions: Other: The same evaluation methods were used for both groups.

INTERVENTIONS:
Other: The same evaluation methods were used for both groups. — No treatment applied to participants and same evaluation methods used in all athletes.

SUMMARY:
The aim of this study was to determine the effect of hamstring muscle length on lunge distance in fencing sword athletes.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of hamstring muscle length on lunge distance in fencing sword athletes. A goniometer was used to assess hamstring muscle length and a tape measure was used to assess lunge distance in 20 athletes who agreed to participate in the study and signed the consent form. We believe that the results of our study will provide new perspectives on increasing the success of fencing sword athletes and reducing their injuries. SPSS 24.0 program will be used for statistical analysis. Pearson correlation test will be applied to evaluate the relationship between hamstring muscle length and lunge distance.

ELIGIBILITY:
Inclusion Criteria:

* Being an active licensed fencing athlete in the Anatolian Archery and Fencing Club
* Being an athlete in the sword branch.
* Being a volunteer to participate in the study
* Being between the ages of 18-30

Exclusion Criteria:

* Having done a strenuous exercise that would affect muscle groups the day before the measurements
* Having used alcohol and/or any medication the day before the measurements

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fencing Sword Branch Athletes
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Hamstring Muscle Length | at baseline
  The athlete was positioned supine with the hip joint at 90 degrees of flexion and was asked to perform active knee extension. The waist and the knee that was not being measured were fixed to the bed. The athlete was asked to slowly extend the knee, and the measurement was recorded with a goniometer at a level where there was no tremor in the knee.
Lunge Distance | at baseline
  Lunge distance was evaluated by measuring the distance between the position of the front foot on the ground in the anguard position and the new position of the front foot on the ground after the lunge, using a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sahin Altac, PT, MSc., Principal Investigator — Halic Üniversity
Locations (1):
- Anatolian Archery and Fencing Club, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gajdosik R, Lusin G. Hamstring muscle tightness. Reliability of an active-knee-extension test. Phys Ther. 1983 Jul;63(7):1085-90. doi: 10.1093/ptj/63.7.1085. PMID 6867117
- See also: ELECTRONIC DEVELOPMENT OF FENCING: A COMPILATION STUDY — http://dergipark.org.tr/tr/download/article-file/602541
- See also: Biomechanics of Lower Extremity Lunge in Fencing — http://dergipark.org.tr/tr/download/article-file/1623878